CLINICAL TRIAL: NCT05572658
Title: mRNA-1345-P901 Study: RSV Outcomes Study Extension
Brief Title: Moderna Vaccine mRNA-1345 Observational Respiratory Syncytial Virus (RSV) Study
Acronym: ROSE
Status: Completed | Type: Observational
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mRNA-1345-P901
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Syncytial Virus
Keywords: Viral Diseases; Messenger RNA; Moderna; mRNA-1345; Effectiveness; Vaccines
MeSH Terms: conditions — Virus Diseases | interventions — mRNA-1345 respiratory syncytial virus vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- mRNA-1345: Exposed: Eligible US participants from the mRNA-1345-P301 (P301) study who received the mRNA-1345 vaccine.
  Interventions: Biological: mRNA-1345
- Placebo/Control: Referent: Eligible US participants from the P301 study who received placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1345 — Sterile liquid for injection
  Groups: mRNA-1345: Exposed
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
  Groups: Placebo/Control: Referent

SUMMARY:
The main goal of this observational study is to describe the health and economic outcomes associated with use of the Moderna mRNA-1345 vaccine.

DETAILED DESCRIPTION:
This study will evaluate real-world data (RWD) and data from eligible United States (US) based participants from Study mRNA-1345-P301 (NCT05127434) for additional health and economic outcomes such as hospitalizations, healthcare resource utilization, disease exacerbations, and costs, associated with usage of the mRNA-1345 vaccine. The results from the current study (mRNA-1345-P901) are intended to complement the results from the mRNA-1345-P301 study. No interventions will be administered during the current study (mRNA-1345-P901).

ELIGIBILITY:
Inclusion Criteria:

P901 inclusion criteria:

* Must be a participant in P301
* Must be based in the US
* Must provide informed consent for P901

P301 key inclusion criteria:

* Adults who are primarily responsible for self-care and activities of daily living.
* Participants may have one or more chronic medical diagnoses (specifically chronic heart failure and chronic obstructive pulmonary disease) but should be medically stable in the opinion of the investigator.
* Body mass index from ≥18 kilograms (kg)/square meter (m^2) to ≤35 kg/m^2.

Exclusion Criteria:

P901 exclusion criteria:

* Receipt of any future licensed RSV vaccine at baseline.
* Receipt of any future licensed RSV vaccines during the study follow-up period will result in censorship on the date the vaccine was received.

All inclusion and exclusion criteria from P301 that are available in the RWD will be applied to the RWD controls, if built.

P301 key exclusion criteria:

* Participation in another clinical research study where participant has received an investigational product (drug/biologic/device) within 45 days before the planned date of the Day 1 vaccination.
* Prior participation in research involving receipt of any investigational RSV product (drug/biologic/device).
* History of a serious reaction to any prior vaccination or Guillain-Barré syndrome within 6 weeks of any prior influenza immunization.
* Received or plans to receive any non-study vaccine within 28 days before or after the Day 1 study injection. The exceptions are seasonal influenza vaccines, pneumococcal vaccines, or authorized or approved vaccines for the prevention of COVID-19 (regardless of type of vaccine), which are not permitted within 14 days before or after the Day 1 study injection. Efforts should be made to space study injection and COVID-19 vaccination by at least 7 and preferably 14 days, but COVID-19 vaccination should not be delayed.

Other inclusion and/or exclusion criteria may apply.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of interest will include P301 participants randomized in the US who provide informed consent and meet eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 10994 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of Hospitalizations for Cardiopulmonary, Cardiovascular, Respiratory, Pneumonia/Influenza, Pneumonia and Complications, or RSV | From Day 15 up to 1 year

SECONDARY OUTCOMES:
Length of Stay of Hospitalizations for Cardiopulmonary, Cardiovascular, Respiratory, Pneumonia/Influenza, Pneumonia and Complications, or RSV | From Day 15 up to 1 year
Mean Total Cost of Hospitalizations and Mean Total Healthcare Cost Related to Cardiopulmonary, Cardiovascular, Respiratory, Pneumonia/Influenza, Pneumonia and Complications, or RSV | From Day 15 up to 1 year
Number of Participants with Use of Mechanical Ventilation, Supplemental Oxygen, and Intensive Care Unit Admissions During Hospitalizations Related to Cardiopulmonary, Cardiovascular, Respiratory, Pneumonia/Influenza, Pneumonia and Complications, or RSV | From Day 15 up to 1 year
Number of Participants with Antibiotic or Corticosteroid Treatment | From Day 15 up to 1 year
Number of Participants with Chronic Obstructive Pulmonary Disease (COPD), Congestive heart failure (CHF), and Asthma | From Day 15 up to 1 year
Number of Participants with First Incidence of Asthma, COPD, and CHF Exacerbations | From Day 15 up to 1 year

CONTACTS AND LOCATIONS:
Locations (109):
- United States (109):
  - Accel Research Site - Achieve - Birmingham - ERN - PPDS, Birmingham, Alabama
  - AES - DRS - Simon Williamson Clinic, PC - Birmingham, Birmingham, Alabama
  - Lakeview Clinical Research, Guntersville, Alabama
  - AES - DRS - Optimal Research Alabama - Huntsville, Huntsville, Alabama
  - Desert Clinical Research, LLC, Mesa, Arizona
  - Hope Research Institute LLC - Phoenix - Hunt - PPDS, Phoenix, Arizona
  - AES - DRS - Phoenix Southeast - Chandler, Phoenix, Arizona
  - AES - DRS - Central Phoenix Medical Clinic, LLC, Phoenix, Arizona
  - Hope Research Institute LLC - Hunt - PPDS, Phoenix, Arizona
  - Hope Research Institute LLC - Hunt - PPDS, Tempe, Arizona
  - Tucson Neuroscience Research - M3 WR, Tucson, Arizona
  - Hope Clinical Research, LLC, Canoga Park, California
  - Velocity Clinical Research - Chula Vista - ERN - PPDS, Chula Vista, California
  - Paradigm Research, La Mesa, California
  - Velocity Clinical Research - Chula Vista - PPDS, La Mesa, California
  - PRI, LLC - Los Alamitos - M3 WR - ERN - PPDS, Los Alamitos, California
  - PRI, LLC - Newport Beach - M3 WR - ERN - PPDS, Newport Beach, California
  - FOMAT Medical Research - FOMAT - HyperCore - PPDS, Oxnard, California
  - Reddy Care Medical, Pomona, California
  - Paradigm Clinical Research Institute Inc - ClinEdge - PPDS, Redding, California
  - Medical Center For Clinical Research - M3 WR - ERN - PPDS, San Diego, California
  - Lynn Institute of Denver - ERN - PPDS, Aurora, Colorado
  - Tekton Research - Fort Collins - Platinum - PPDS, Fort Collins, Colorado
  - Tekton Research - Longmont - Platinum - PPDS, Longmont, Colorado
  - Paradigm Clinical Research Institute Inc - ClinEdge - PPDS, Wheat Ridge, Colorado
  - Velocity Clinical Research - New Smyrna Beach - ERN - PPDS, Edgewater, Florida
  - Fleming Island Center For Clinical Research - ERN-PPDS, Fleming Island, Florida
  - Velocity Clinical Research - Hallandale Beach - ERN - PPDS, Hallandale, Florida
  - Jacksonville Center For Clinical Research - ERN - PPDS, Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Multi-Specialty Research Associates, Inc. M3 WR, Lake City, Florida
  - Accel Research Sites - Maitland - ERN - PPDS, Maitland, Florida
  - AES - DRS - Synexus Clinical Research US, Inc. - St. Petersburg, Pinellas Park, Florida
  - AES - DRS - Synexus Clinical Research US, Inc. - The Villages, The Villages, Florida
  - Palm Beach Research - ClinEdge - PPDS, West Palm Beach, Florida
  - Clinical Site Partners - Winter Park - HyperCore - PPDS, Winter Park, Florida
  - Masters of Clinical Research Inc., Augusta, Georgia
  - Centricity Research - Roswell - HyperCore - PPDS, Columbus, Georgia
  - IResearch Atlanta LLC - ClinEdge - PPDS, Decatur, Georgia
  - Javara, Inc./Privia Medical Group Georgia, LLC - Fayetteville - Javara - PPDS, Fayetteville, Georgia
  - Mount Vernon Clinical Research, LLC - M3 WR - ERN - PPDS, Sandy Springs, Georgia
  - Meridian Clinical Research (Savannah Georgia) - Platinum - PPDS, Savannah, Georgia
  - Clinical Research Atlanta - ERN-PPDS, Stockbridge, Georgia
  - Velocity Clinical Research - Boise - PPDS, Meridian, Idaho
  - AES - DRS - Synexus Clinical Research US, Inc. - Chicago, Chicago, Illinois
  - Affinity Health (Oak Brook), Oak Brook, Illinois
  - DM Clinical Research - Chicago - ERN - PPDS, River Forest, Illinois
  - AES - DRS - Synexus Clinical Research US, Inc. - Evansville, Evansville, Indiana
  - Velocity Clinical Research - Valparaiso - ERN - PPDS, Valparaiso, Indiana
  - Versailles Family Medicine, PLLC, Versailles, Kentucky
  - Meridian Clinical Research (Baton Rouge-Louisiana) - Platinum - PPDS, Baton Rouge, Louisiana
  - Benchmark Research - Covington - HyperCore - PPDS, Covington, Louisiana
  - Benchmark Research - Metairie - HyperCore - PPDS, Metairie, Louisiana
  - Clinical Trials of America, LLC, Monroe, Louisiana
  - DelRicht Clinical Research, LLC - Internal - Covington - PPDS, New Orleans, Louisiana
  - Javara Research Inc. - Annapolis - Javara - PPDS, Annapolis, Maryland
  - CBH Health - CenExcel CBH - PPDS, Gaithersburg, Maryland
  - Meridian Clinical Research (Rockville Maryland) - Platinum - PPDS, Rockville, Maryland
  - Great Lakes Research Institute, Southfield, Michigan
  - DM Clinical Research - Southfield - ERN - PPDS, Southfield, Michigan
  - Clinical Research Institute, Inc - CRN - PPDS, Plymouth, Minnesota
  - AES - DRS - Synexus Clinical Research US, Inc. - Minneapolis, Richfield, Minnesota
  - AES - DRS - Synexus Clinical Research US, Inc. - St. Louis, St Louis, Missouri
  - Montana Medical Research, Missoula, Montana
  - Skyline Medical Center, PC, Elkhorn, Nebraska
  - Methodist Physicians Clinic - Prairie - CCT Research, Fremont, Nebraska
  - Meridian Clinical Research (Grand Island) - Platinum - PPDS, Grand Island, Nebraska
  - Meridian Clinical Research (Omaha-Nebraska) - Platinum - PPDS, Omaha, Nebraska
  - Meridian Clinical Research, LLC (Lincoln Nebraska) - Platinum - PPDS, Omaha, Nebraska
  - CCT Research, Papillion, Nebraska
  - HEALOR Primary Care - Physicians Las Vegas, Las Vegas, Nevada
  - Excel Clinical Research - Las Vegas, Las Vegas, Nevada
  - Velocity Clinical Research - East Syracuse - ERN - PPDS, East Syracuse, New York
  - Meridian Clinical Research (Endwell-New York) - Platinum - PPDS, Endwell, New York
  - Meridian Clinical Research (Dakota Dunes-South Dakota) - Platinum - PPDS, Endwell, New York
  - Drug Trials America, Hartsdale, New York
  - AES - DRS - Synexus Clinical Research US, Inc. - New York, New York, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Carolina Institute for Clinical Research - M3 WR - ERN - PPDS, Fayetteville, North Carolina
  - Velocity Clinical Research - Cincinnati - ERN - PPDS, Blue Ash, Ohio
  - Meridian Clinical Research - Cincinnati - Platinum - PPDS, Cincinnati, Ohio
  - CTI Clinical Research Center - PPDS, Cincinnati, Ohio
  - AES - DRS - Synexus Clinical Research US, Inc. - Cincinnati, Cincinnati, Ohio
  - Tekton Research - Oklahoma - Platinum - PPDS, Yukon, Oklahoma
  - Tekton Research Inc., Yukon, Oklahoma
  - Hatboro Medical Associates PC, Hatboro, Pennsylvania
  - DM Clinical Research - Philadelphia - ERN - PPDS, Philadelphia, Pennsylvania
  - Tekton Research Inc., Austin, Texas
  - PanAmerican Clinical Research LLC, Brownsville, Texas
  - Family Medicine Associates of Texas - Hunt - PPDS, Carrollton, Texas
  - Javara, Inc./Texas Health Care, PLLC (d/b/a/ Privia Medical Group - North Texas) - Javara - PPDS, Fort Worth, Texas
  - Allure Health LLC, Friendswood, Texas
  - Village Health Partners Frisco Medical Village, Frisco, Texas
  - DM Clinical Research - Texas Center For Drug Development - ERN - PPDS, Houston, Texas
  - DM Clinical Research - Texas Center for Drug Development - Humble - ERN - PPDS, Humble, Texas
  - Ventavia Research Group - Platinum - PPDS, Keller, Texas
  - AIM Trials, Plano, Texas
  - Clinical Trials of Texas, Inc. - PPDS, San Antonio, Texas
  - Javara, Inc./Texas Health Care, PLLC (d/b/a/ Privia Medical Group - North Texas) - Stephenville - Ja, Stephenville, Texas
  - DM Clinical Research - Sugarland - ERN - PPDS, Sugar Land, Texas
  - DM Clinical Research - ERN, Tomball, Texas
  - DM Clinical Research - ERN - PPDS, Tomball, Texas
  - Cope Family Medicine - Ogden Clinic - CCT, Bountiful, Utah
  - Olympus Family Medicine - CCT Research, Holladay, Utah
  - South Ogden Family Medicine/Ogden Clinic - CCT Research, South Ogden, Utah
  - Velocity Clinical Research - Banning - ERN - PPDS, West Jordan, Utah
  - Meridian Clinical Research - Family Practice Ports - Portsmouth - Platinum - PPDS, Portsmouth, Virginia
  - Rainier Clinical Research Center, Renton, Washington
  - Seattle Womens: Health, Research, Gynecology, Seattle, Washington